CLINICAL TRIAL: NCT04137978
Title: Open Label, Multicentre Study, Evaluating the Safety, Tolerability, Efficacy, Compliance and Acceptability of Alkalising Treatments at Long-term in Patients With Cystinuria
Brief Title: Study Evaluating Patients With Cystinuria
Status: Withdrawn | Phase: Phase 2 / Phase 3 | Type: Interventional
Why Stopped: Unspecified business decision/strategic reason
Sponsor: Advicenne Pharma (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: B14CS
Record Dates: First submitted 2019-10-18; First posted 2019-10-24 (Actual); Last update posted 2024-03-12 (Actual); Status verified 2024-03

CONDITIONS: Cystinuria
MeSH Terms: conditions — Cystinuria | interventions — Potassium Citrate; potassium bicarbonate; Standard of Care

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- ADV7103 (Active Comparator): Patients receive ADV7103 twice a day at optimal dose. Each dose of ADV7103 contains a fixed ratio of 1/3 of ADV7103-CK (potassium citrate) and 2/3 of ADV7103-BK (potassium bicarbonate) based on the mass of active substances.
  Other Names:
  • Potassium Citrate and Potassium Bicarbonate
  Interventions: Drug: ADV7103
- Standard of care comparator (Active Comparator): Alkalinising treatment (SoC) taken at the usual dose and frequency
  Interventions: Drug: Standard of Care

INTERVENTIONS:
Drug: ADV7103 — Patients receive ADV7103 twice a day at optimal dose.
  Other Names: Potassium Citrate and Potassium Bicarbonate
  Arms: ADV7103
Drug: Standard of Care — Cohort of patients with cystinuria, matching-pair for age category to the patients of ADV7103 Cohort, will receive their own alkalinising treatment (SoC) taken at the usual dose and frequency and will follow their usual first intention treatment (hydration and diet) for a 2-year-period.
  Arms: Standard of care comparator

SUMMARY:
This is an open label, multicentre study, evaluating the safety, tolerability, efficacy, compliance and acceptability of alkalising treatments at long-term in patients with cystinuria.

DETAILED DESCRIPTION:
B14CS study is an extension study which follows the B12CS-B13CS study. Patients who have participated in B12CS-B13CS Study will have the possibility to switch to B14CS Study for a long-term treatment period (2 year-period).

The B14CS Study is an open-label long-term study and including 2 types of cohorts.

* ADV7103 Cohort: Cohort of patients who will have completed either B12CS or B13CS Study. Following an optional titration period (for B12CS Study subjects), all patients will be maintained at their ADV7103 optimal dose for a 2-year-period.
* SoC Cohort: Cohort of patients with cystinuria, matching-pair for age category to the patients of ADV7103 Cohort, will receive their own alkalinising treatment (SoC) taken at the usual dose and frequency and will follow their usual first intention treatment (hydration and diet) for a 2-year-period. This cohort is designed in order to contextualize the safety, tolerability and efficacy of the long-term ADV7103 treatment.

The B14CS Study will be composed of 3 periods (more detailed hereafter):

* Lead-in Period: Period of 3 weeks, during which the treatment (ADV7103 or SoC) will be taken at the optimal dose as previously defined (Maintenance Phase). The Lead-in Period can include a Titration Phase, for ADV7103 B12CS Cohort only, in order to define the individual optimal dose of ADV7103 for the patients of this cohort;
* Assessment Period: Period of 7 days to evaluate the effect of study products (ADV7103 and SoC) at the optimal dose;
* Follow-up Period: Period of 23 months to evaluate the effects of the study products (ADV7103 and SoC) at long-term.

ELIGIBILITY:
Inclusion Criteria:

* For ADV7103 cohort:

  1. Patient who has participated to and completed the previous B12CS Study or B13CS Study.
  2. Patient for whom the safety and tolerability of ADV7103 were satisfactory during B12CS Study or B13CS Study.
  3. Female patient of childbearing potential (defined by the Clinical Trial Facilitation Group (CTFG) as woman fertile, following menarche until becoming post-menopausal unless permanently sterile*) using an acceptable effective birth control method** and having a negative pregnancy test at the inclusion, or a woman postmenopausal*** or a woman surgically sterilized*.
  4. Patient and/or parents or legal representative(s) who is(are) willing and able to participate in the study, to understand and to comply with study procedures for the entire length of the study.
  5. Patient or parents or legal representative(s) who has(have) provided a signed written informed consent.
  6. Patient of ≤17 Patient of ≤17 years of age for whom the assent has been collected or has been tried to be collected.
  7. Patient who is affiliated to a social health insurance system and/or in compliance with the recommendations of the national law in force relating to biomedical research.

For Standard of Care cohort:

1. Patient who has a diagnosis of cystinuria based on medical diagnosis (at least one previous or current episode of calculus of cystine, and/or one previous or current episode of cystine crystalluria) or on genetic diagnosis (only for patients of Subset 4).
2. Patient treated with an alkalising treatment at a well-adapted dose (defined as a daily dose deemed by the investigator aiming to maintain overtime urinary pH value ≥ 7.0 and/or compatible with an acceptable safety profile and/or patient's constraints or compliance).
3. Patient male or female, including child aged between 6 months and 17 years old and adult aged ≥ 18 years old up to 70 years old.
4. Female patient of childbearing potential (defined by the Clinical Trial Facilitation Group (CTFG) as woman fertile, following menarche until becoming post-menopausal unless permanently sterile*) using an acceptable effective birth control method** and having a negative pregnancy test at the inclusion, or a woman postmenopausal*** or a woman surgically sterilized*.
5. Patient and/or parents or legal representative(s) who is(are) willing and able to participate in the study, to understand and to comply with study procedures for the entire length of the study.
6. Patient or parents or legal representative(s) who has/have provided a signed written informed consent.
7. Patient of ≤17 years of age for whom the assent has been collected or has been tried to be collected.
8. Patient who is affiliated to a social health insurance system and/or in compliance with the recommendations of the national law in force relating to biomedical research.

Exclusion Criteria:

* For ADV7103 cohort:

  1. Patient who has not participated to B12CS study or B13CS study
  2. Patient for whom any safety issue could contraindicate her/his participation to the extension study

For Standard of Care cohort:

1. Patient that is receiving the second line therapy -- cystine chelating agents (sulfhydryl compounds).
2. Patient who presents kalaemia > 5.0 mmol/L.
3. Patient who presents a moderate or severe renal impairment (estimated glomerular filtration rate (eGFR) < 45 mL/min/1.73 m2 according to Schwartz formula for the children and both MDRDs and CKD-EPI for adults).
4. Patient who presents - barring the study disease - any previous or concurrent medical condition or any laboratory or clinical findings or any other condition that in the opinion of the investigator would be negatively affected by the study product or that would affect the study product or that precludes his participation, e.g. uncontrolled diabetes mellitus, adrenal insufficiency, cardiac impairment, repeated infections, metabolic alkalosis, chronic diarrhoea.
5. Female patient who is pregnant or breast-feeding.
6. Patient who cannot stop potassium sparing diuretics (e.g. antagonists of aldosterone as such spironolactone, canrenoate and eplerenone, amiloride, triamterene), angiotensin converting enzyme inhibitors, angiotensin II receptor antagonists, tacrolimus, potassium desodic salts.
7. Patient who received any medication that could interfere with the study treatment within 4 weeks before the inclusion in the study, including angiotensin converting enzyme inhibitors, angiotensin II receptor antagonists, tacrolimus, potassium desodic salts, antibiotics.
8. Patient who received potassium sparing diuretics 6 weeks before the inclusion in the study.
9. Patient who is admitted to hospital in emergency settings.
10. Patient who participated in a clinical trial within the last 3 months before enrolment.
11. Patient who is at risk of non-compliance in the judgment of the investigator.
12. Patient who could present any other condition, which in the opinion of the investigator, would preclude participation in the study.
13. Patient who cannot be contacted in case of emergency.
14. Patient under any administrative or legal supervision.

Ages: 6 Months to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2024-05-01 (Estimated); Primary Completion 2025-06 (Estimated); Study Completion 2025-08 (Estimated)

PRIMARY OUTCOMES:
Percentage of urinary pH values ≥ 7.0 during 24h on Day 7 (after ADV7103 treatment period) | 7 Days
  To evaluate the safety and the tolerability of ADV7103 and standard of care (SoC) after a long-term treatment.

CONTACTS AND LOCATIONS:
Overall Officials: Luc-André Granier, M.D., Study Director — Advicenne Pharma
Locations (13):
- Belgium (2):
  - Cliniques Universitaires Saint-Luc, Brussels
  - UZ Leuven, Gasthuisberg Hospital, Leuven
- France (11):
  - CHU de Bordeaux - Hôpital Pellegrin, Bordeaux
  - Centre Hospitalier Universitaire de Lyon, Bron
  - CHU Grenoble, Grenoble
  - CHRU Lille, Lille
  - CHU Pitié-Salpétrière, Paris
  - Hôpital Necker AP-HP, Paris
  - Hôpital Necker Enfants Malades, Paris
  - Hôpital Ténon - Explorations fonctionnelles Mutlidisciplinaires et INSERM UMR S 1155, Paris
  - Hôpital Américain CHU de Reims, Reims
  - CHU Reims, Reims
  - CHU Purpan, Toulouse

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Company website — http://advicenne.com